CLINICAL TRIAL: NCT00139763
Title: A US Randomized Questionnaire-Based Trial Assessing The Impact Of The Availability Of Inhaled Insulin On Therapeutic Choice In Patients With Suboptimally Controlled Type 2 Diabetes
Brief Title: US Inhaled Insulin Therapeutic Choice Questionnaire Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: A2171066
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Procedure: Educational Materials

SUMMARY:
This is a questionnaire based study (no study drug is involved) that asks if more patients with uncontrolled type 2 diabetes on diabetes pills will choose insulin as the next treatment choice if inhaled insulin were available in addition to all currently available treatments, compared with if inhaled insulin was not available as part of currently available treatments.

This study will also ask if patients with uncontrolled type 2 diabetes currently managed on diabetes pills + once daily insulin will choose as the next treatment choice to take insulin multiple times a day if inhaled insulin were available in addition to all currently available treatments, compared with if inhaled insulin was not available as part of currently available treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, age > = 18 years and <= 80 years with a diagnosis of type 2 diabetes made at least 6 months prior to study entry
* Currently treated with either:
* 2 or more oral antidiabetic agents, OR 1 or more oral antidiabetic agents and insulin glargine

Exclusion Criteria:

* Type 1 diabetes
* Smoking within the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740
Dates: Start 2005-07; Study Completion 2006-03

PRIMARY OUTCOMES:
Will availability of inhaled insulin result in more type 2 diabetes patients choosing a treatment that involves insulin (if now on >2 OAs) or a more intensive insulin regimen (if now on OAs + glargine) compared to only standard therapies available

SECONDARY OUTCOMES:
Determine both patient and MD reasons for treatment choices made. Determine if treatment choice is influenced by physician specialty or patient ethnicity. Determine how cost impacts patient treatment choice.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (39):
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tempe, Arizona
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Hayden, Idaho
  - Pfizer Investigational Site, Nampa, Idaho
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Elkton, Maryland
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Margate City, New Jersey
  - Pfizer Investigational Site, Santa Fe, New Mexico
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Morehead City, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Statesville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Orangeburg, South Carolina
  - Pfizer Investigational Site, Simpsonville, South Carolina
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Madisonville, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Bennington, Vermont
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171066&StudyName=US+Inhaled+Insulin+Therapeutic+Choice+Questionnaire+Study